CLINICAL TRIAL: NCT06771089
Title: A Comparative Study of the Effectiveness of a Therapeutic Exercise Protocol Vs a Mobilisation with Movement Protocol in Improving Ankle Dorsiflexion in Amateur Football Players. Randomised Controlled Pilot Study
Brief Title: Effectiveness of a Therapeutic Exercise Protocol Vs a Mobilisation with Movement Protocol in Improving Ankle Dorsiflexion in Amateur Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Iris Machado de Oliveira (Unknown); Aldara Vázquez Méndez (Unknown); Adrian Eiró Fernández (Unknown)
Responsible Party: Principal Investigator, Irimia Mollinedo Cardalda, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205-2024-1
Record Dates: First submitted 2024-12-30; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Ankle Dorsiflexion
Keywords: Ankle dorsiflexion; Football; Therapeutic exercise; Mobilization with movement; Knee dynamic valgus
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manual therapy group (MTG) (Experimental): The MTG group received an intervention based on anterior-posterior mobilizations of the talus and fibula and taping, both based on Mulligan® techniques.
  Interventions: Other: Manual therapy and bandaging
- Therapeutic exercise group (EG) (Experimental): The EG group underwent a therapeutic exercise protocol lasting approximately 5-10 minutes, performed before regular training sessions.
  Interventions: Other: Therapeutic exercise
- Control group (CG) (Placebo Comparator): The CG group received no specific treatment; they only participated in the current training sessions.
  Interventions: Other: No specific treatment

INTERVENTIONS:
Other: Manual therapy and bandaging — The MTG group received an intervention based on anterior-posterior mobilizations of the talus and fibula and taping, both based on Mulligan® techniques Individually, participants received Grade IV passive mobilizations lasting approximately 30 seconds, totalling 12 active mobilizations performed by the participant. Furthermore, a tape was applied, placed on the anterior part of the talus with a posterior and caudal direction, with its ends anchored near the heel. Due to its placement, this taping maintained a sustained posterior force on the talus throughout the training session. This intervention was conducted on the affected limb(s) with DF deficits.
  Arms: Manual therapy group (MTG)
Other: Therapeutic exercise — Therapeutic exercise protocol lasting approximately 5-10 minutes, performed before regular training sessions. It included 2 exercises, each performed in 3 sets of 10 repetitions with 1-minute rest intervals.
  Exercise 1: Weighted DF in a kneeling position. From this position, ankle DF is performed with the front leg, on which the weight of the arms and the torso is placed to force the movement.
  Exercise 2: Ankle lunge with band resistance at the ankle. The player performs ankle DF with a medium-resistance green Theraband® providing a posterior force vector on the talus.
  This intervention was applied to the affected limb(s) with ankle DF limitations and was supervised by a physiotherapist. It was performed before training session at each club's facilities.
  Arms: Therapeutic exercise group (EG)
Other: No specific treatment — The Control group received no specific treatment; they only participated in the current training sessions.
  Arms: Control group (CG)

SUMMARY:
Objective: To evaluate and compare the immediate and short-term effectiveness of a therapeutic exercise protocol and a mobilisation with movement protocol, compared with a control group, in improving ankle dorsiflexion in amateur footballers.

Material and methods: A single-blind randomised controlled pilot study was developed. Participants were amateur football players randomized into 3 groups (therapeutic exercise, mobilization with movement and control). The intervention was carried out with 2 weekly sessions for 4 weeks. Assessment tools included the Ankle Lunge Test and the Single Leg Squat.

ELIGIBILITY:
Inclusion Criteria:

* Football players over 18 years old who train a minimum of 3 days a week.
* Football players with ankle DF less than 9 cm or a difference greater than 1.5 cm between both feet, measured with the Ankle Lunge Test (ALT) using the LegMOtion© device.

Exclusion Criteria:

* Players who, during the ALT, achieve less than 9 cm or a difference greater than 1.5 cm between both feet but reporting limitation due to tension in the gastrocnemius muscle.
* Those with serious traumatic or rheumatological conditions that may interfere with the study.
* Players who have participated in specific programs to improve ankle DF in the last 3 months.
* Players with a history of ankle-foot surgery within the last 6 months.
* Non-registered players training in those clubs.
* Players unable to arrive 20 minutes prior to the beginning of the training session.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Ankle dorsiflexion with Ankle Lunge Test (ALT) using the LegMOtion© device. | 4 weeks
  ALT: ankle DF was measured in cm. The player stands with the foot to be assessed placed behind a black line on the device, while the other foot remains on the floor behind the tested foot. The player attempts to touch a metal rod with the knee without lifting the heel off the floor. The rod's position is adjusted to the maximum distance reached with difficulty. 3 repetitions were carried out and an average of the 3 repetitions was calculated to obtain the maximum ankle DF measurement. Both feet were measured.

SECONDARY OUTCOMES:
Dynamic knee valgus with the Single Leg Squat (SLS) test. | 4 weeks
  SLS: The participant, barefoot on a firm, flat surface, first performed 2 practice SLS repetitions unmeasured., then 2 consecutive sets of 5 repetitions were evaluated and the worst set was chosen for analysis., allowing for speed and compensation adjustments as fatigue developed. Each limb was tested. The examiner, positioned directly in front of the participant, recorded the activity with a mobile device. Movement execution was analysed using the Kinovea© software, with analysis focused on measuring the Q angle for each repetition, selecting the largest angle from the 5 executions for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vigo, Pontevedra, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided